CLINICAL TRIAL: NCT01274299
Title: Facial Dimensions in Infants and Toddlers
Brief Title: Measurements of Facial Dimensions in Infants and Toddlers 0-4 Years of Age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Israel Amirav, Ziv Medical Center
Other Study IDs: 0067-10-ZIV
Record Dates: First submitted 2010-12-28; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Infant Development
Keywords: Infants; morphometry; face; 3D
MeSH Terms: conditions — Facies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants: Healthy 0-4 years of age both boys and girls
  Interventions: Procedure: Digital camera picture

INTERVENTIONS:
Procedure: Digital camera picture — A digital camera will be used to take a 3D picture the face of each infant. Off line measurements of landmarks on the face will be marked and dimensions will be calculated using a special analysis software.
  Other Names: none applicable

SUMMARY:
Anthropometric data of infants' face will be obtained using special 3D scanners and software.

DETAILED DESCRIPTION:
A digital camera will be used to take a 3D picture the face of each infant. Off line measurements of landmarks on the face will be marked and dimensions will be calculated using a special analysis software.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants, 0-4 years of age

Exclusion Criteria:

* Facial anomalies

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-11; Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Facial Dimensions | 5 minutes
  Landmarks that are relevant to face mask application such as the distance from the chin to the bridge of the nose will be marked and measured.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Amirav, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical center, Safed, Israel

REFERENCES:
- [Derived] Amirav I, Luder AS, Halamish A, Marzuk C, Daitzchman M, Newhouse MT. Computerized Dead-Space Volume Measurement of Face Masks Applied to Simulated Faces. Respir Care. 2015 Sep;60(9):1247-51. doi: 10.4187/respcare.03813. Epub 2015 May 5. PMID 25944944
- [Derived] Amirav I, Luder AS, Halamish A, Raviv D, Kimmel R, Waisman D, Newhouse MT. Design of aerosol face masks for children using computerized 3D face analysis. J Aerosol Med Pulm Drug Deliv. 2014 Aug;27(4):272-8. doi: 10.1089/jamp.2013.1069. Epub 2013 Sep 28. PMID 24074142